CLINICAL TRIAL: NCT01162551
Title: Phase 2 Trial of Sirolimus and Methotrexate in Relapsed/Refractory Lymphoblastic Leukemia and Lymphoma
Brief Title: Trial of Sirolimus and Methotrexate in Relapsed/Refractory Lymphoblastic Leukemia and Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-007444; 6137-09 (Other Grant/Funding Number: Leukemia and Lymphoma Society)
Record Dates: First submitted 2010-06-25; First posted 2010-07-14 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Cancer; Leukemia; Lymphoma
Keywords: Leukemia; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Neoplasms; Leukemia; Lymphoma; Lymphoma, Non-Hodgkin | interventions — Sirolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus and Methotrexate (Experimental): Sirolimus: Oral bolus on day 1, then daily oral dose days 2-28. Dose will be altered to maintain a sirolimus trough level between ≥ 8 and ≤ 13. Trough levels will be checked weekly.
  Methotrexate: Oral 20 mg/m2/week on Days 2, 9, 16, 23.
  One cycle is 28 days
  Interventions: Drug: Sirolimus and Methotrexate

INTERVENTIONS:
Drug: Sirolimus and Methotrexate — Single Arm Efficacy Trial:
  Sirolimus: Oral bolus on day 1, then daily oral dose days 2-28. Dose will be altered to maintain a sirolimus trough level between ≥ 8 and ≤ 13. Trough levels will be checked weekly.
  Methotrexate: Oral 20 mg/m2/week on Days 2, 9, 16, 23.
  One cycle is 28 days.
  Other Names: SIROLIMUS; AY-22989; rapamycin; Rapamune®; METHOTREXATE; MTX; amethopterin; Trexall®

SUMMARY:
This is a phase 2 study looking at efficacy and toxicity of oral sirolimus in combination with oral methotrexate in children with refractory/relapsed ALL or NHL.

Secondary objectives include characterizing the trough levels produced by administration of oral sirolimus in children with refractory/relapsed ALL/NHL and to evaluate the effect of sirolimus on intracellular targets related to mTOR inhibition.

DETAILED DESCRIPTION:
At present children who have bone marrow or combined bone marrow and extramedullary relapses of acute leukemia while on therapy have 5-20% of long-term survival. Newer, targeted agents need to be identified and integrated into the present cytotoxic chemotherapy regimens. Biologically targeted cancer agents, including signal transduction inhibitors like mammalian target of rapamycin inhibitors (MTIs), have shown great promise in treating hematologic malignancies. A Phase 1 trial of sirolimus (an MTI) alone performed at CHOP has been well tolerated with no DLTs and has evidence of hitting the biologic target. While signal transduction inhibitors may be efficacious as single agents, it is more likely that these targeted agents will demonstrate greater efficacy in combination with other cytotoxic agents.Based upon pre-clinical humanized ALL mouse models we propose to study the toxicity and efficacy of adding sirolimus to oral methotrexate in relapsed and refractory patients.

Patients < 25 years of age, at time of enrollment, with second or greater relapse of ALL or NHL (lymphoblastic lymphoma or peripheral T-cell lymphoma) are eligible. ALL patients must have at least 10% blasts in their marrow and NHL patients must have radiologic or physical evidence of recurrence.

Patients will be started on daily oral sirolimus that is dosed based upon goal trough levels and weekly oral methotrexate. All therapy can be done as an outpatient.

ELIGIBILITY:
Inclusion Criteria:

* Patients </= 25 years of age, at time of enrollment, with second or greater relapse of ALL or NHL. For ALL must have histologic diagnosis with >10% blasts in the marrow and for lymphoblastic lymphoma or peripheral T-cell lymphoma must have radiologic or physical evidence of recurrence.
* Lansky > 50% or Karnofsky > 50%
* Negative Pregnancy Test
* Creatinine clearance or radioisotope GFR > 70ml/min/m2 OR serum creatinine based on age /gender
* Pulse ox >94%
* Total Bilirubin <1.5 x normal for age
* ALT < 5 x normal for age
* Albumin > 2g/dL
* Shortening fraction by echo > 28% OR ejection fraction > 50% by gated radionuclide study

Exclusion Criteria:

* Patient has known allergies to sirolimus,FK-506 or mTOR inhibitors
* Patient is taking other investigational anti-neoplastic drugs
* Patient received no myelosuppressive chemo within 14 days
* < 14 days have elapsed since local palliative XRT (small port) < 28 days since prior craniospinal XRT or 50% radiation of pelvis <28 days if other substantial BM radiation
* Hematopoietic growth factors within 7 days of entry (except erythropoietin.)
* Patient has taken any biologic agents within 14 days
* Post BMT/SCT - evidence of active GVHD, at least > 3 months must have elapsed
* Patient has uncontrolled infection (if patients with fungal disease, stable for < 14 days and patients with bacteremia without negative blood culture
* Existing non-hematologic toxicities > grade 2

Use of steroids or hydroxyurea is permitted upto 14 days prior to entry.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2010-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan R. Rheingold, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Teachey DT, Sheen C, Hall J, Ryan T, Brown VI, Fish J, Reid GS, Seif AE, Norris R, Chang YJ, Carroll M, Grupp SA. mTOR inhibitors are synergistic with methotrexate: an effective combination to treat acute lymphoblastic leukemia. Blood. 2008 Sep 1;112(5):2020-3. doi: 10.1182/blood-2008-02-137141. Epub 2008 Jun 10. PMID 18544682
- [Background] Houghton PJ, Morton CL, Kolb EA, Gorlick R, Lock R, Carol H, Reynolds CP, Maris JM, Keir ST, Billups CA, Smith MA. Initial testing (stage 1) of the mTOR inhibitor rapamycin by the pediatric preclinical testing program. Pediatr Blood Cancer. 2008 Apr;50(4):799-805. doi: 10.1002/pbc.21296. PMID 17635004
- [Background] Teachey DT, Obzut DA, Cooperman J, Fang J, Carroll M, Choi JK, Houghton PJ, Brown VI, Grupp SA. The mTOR inhibitor CCI-779 induces apoptosis and inhibits growth in preclinical models of primary adult human ALL. Blood. 2006 Feb 1;107(3):1149-55. doi: 10.1182/blood-2005-05-1935. Epub 2005 Sep 29. PMID 16195324
- [Background] Brown VI, Fang J, Alcorn K, Barr R, Kim JM, Wasserman R, Grupp SA. Rapamycin is active against B-precursor leukemia in vitro and in vivo, an effect that is modulated by IL-7-mediated signaling. Proc Natl Acad Sci U S A. 2003 Dec 9;100(25):15113-8. doi: 10.1073/pnas.2436348100. Epub 2003 Dec 1. PMID 14657335
- [Background] Luger S, Perl A, Kemner A. A phase I dose escalation study of the mTOR inhibitor sirolimus and MEC chemotherapy targeting signal transduction in leukemic stem cells for acute myeloid leukemia. . Blood. 2006;106:161.
- [Background] Morrison DJ, Hogan LE, Condos G, Bhatla T, Germino N, Moskowitz NP, Lee L, Bhojwani D, Horton TM, Belitskaya-Levy I, Greenberger LM, Horak ID, Grupp SA, Teachey DT, Raetz EA, Carroll WL. Endogenous knockdown of survivin improves chemotherapeutic response in ALL models. Leukemia. 2012 Feb;26(2):271-9. doi: 10.1038/leu.2011.199. Epub 2011 Aug 16. PMID 21844871
- [Background] Sheen C, Vincent T, Barrett D, Horwitz EM, Hulitt J, Strong E, Grupp SA, Teachey DT. Statins are active in acute lymphoblastic leukaemia (ALL): a therapy that may treat ALL and prevent avascular necrosis. Br J Haematol. 2011 Nov;155(3):403-7. doi: 10.1111/j.1365-2141.2011.08696.x. Epub 2011 May 9. No abstract available. PMID 21554258
- [Background] Barrett D, Brown VI, Grupp SA, Teachey DT. Targeting the PI3K/AKT/mTOR signaling axis in children with hematologic malignancies. Paediatr Drugs. 2012 Oct 1;14(5):299-316. doi: 10.2165/11594740-000000000-00000. PMID 22845486

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus and Methotrexate: Sirolimus: Oral bolus on day 1, then daily oral dose days 2-28. Dose will be altered to maintain a sirolimus trough level between ≥ 8 and ≤ 13. Trough levels will be checked weekly.
  Methotrexate: Oral 20 mg/m2/week on Days 2, 9, 16, 23.
  One cycle is 28 days
  Sirolimus and Methotrexate: Single Arm Efficacy Trial:
  Sirolimus: Oral bolus on day 1, then daily oral dose days 2-28. Dose will be altered to maintain a sirolimus trough level between ≥ 8 and ≤ 13. Trough levels will be checked weekly.
  Methotrexate: Oral 20 mg/m2/week on Days 2, 9, 16, 23.
  One cycle is 28 days.
Period: Overall Study
Arm/Group | Sirolimus and Methotrexate
Started | 3 (2 subjects were enrolled but withdrew before receiving any study treatment)
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There were 5 participants enrolled, their data is included in the participant flow and demographic section. 2 of these subjects withdrew before staring therapy and are not included in the outcome measures or in adverse event analysis.
Arm/Group | Sirolimus and Methotrexate
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 12 [7 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Number of participants who achieve a Complete Response (CR), Complete Response with in the absence of total platelet recovery (CRp), or Partial Response (PR). Per response criteria in this protocol: Complete Response (CR) - M1 bone marrow (<5% blasts) with no evidence of circulating blasts or extramedullary disease and recovery of peripheral blood counts (absolute neutrophil count (ANC)> 500/μL and platelets > 50,000/ μL); Complete Response in the absence of total platelet recovery (CRp) - M1 bone marrow (<5% blasts) with no evidence of circulating blasts or extramedullary disease with recovery of peripheral blood counts except for platelets (ANC> 500/μL, platelets < 50,000uL); and Partial Response (PR) - M2 bone marrow (5% but <25% blasts), with no evidence of circulating blasts or extramedullary disease and normalization of peripheral blood counts (ANC > 500/μL and platelets >50,000/μL).
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | Sirolimus and Methotrexate
Number analyzed (Participants) | 3
participants
  CR | 0
  CRp | 0
  PR | 0

2. Secondary Outcome: Number of Dose Adjustments To Maintain Trough Levels
Description: One goal of this study is to maintain trough levels of sirolimus within a certain range. The outcome measure counts the number of dose adjustments up or down that were needed to meet goal level based on weekly tough level measurements.
Time Frame: Day 28
Population: 3 patients had weekly sirolimus levels analyzed.
Measure: Number; unit: Dose level adjustments
Units Other Than Participants: blood samples
Arm/Group | Sirolimus and Methotrexate
Number analyzed (Participants) | 3
Number analyzed (blood samples) | 9
Dose level adjustments
  Dose level increase | 2
  Dose level decrease | 1

ADVERSE EVENTS:
Time Frame: 4.5 years
Arm/Group | Sirolimus and Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus and Methotrexate (N=3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Increased work of breathing requiring CPAP. Due to disease progression and abdominal competition from increasing HSM
Hematuria (Renal and urinary disorders) | 1 (1) — Hematuria due to BK virus, unrelated
torsades (Cardiac disorders) | 1 (1) — Torsade due to hypokalemia and hypophosphatemia. Combined with Zofran had prolonged QTC
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus and Methotrexate (N=3)
Cytopenias (Blood and lymphatic system disorders) | 2 (2)
electrolyte abnormalitles (Metabolism and nutrition disorders) | 2 (2)
fever (General disorders) | 1 (1) — Fever, febrile neutropenia, bacteremia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-02-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT01162551/Prot_SAP_000.pdf